CLINICAL TRIAL: NCT02489149
Title: Food and Nutrition Education in Quilombolas Communities With Food Insecurity: Intervention Based on Traditional Food Practices, Healthy Eating Promotion and Enforceability of Human Right to Adequate Food
Brief Title: Food and Nutrition Education in Quilombolas Communities With Food Insecurity: Multi-sector Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Principal Investigator, Marilda Borges Neutzling, Professor, Federal University of Rio Grande do Sul
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25445
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: food insecurity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-sector interventions (Experimental): Multi-sector interventions
  * Multi-sector interventions to enhance food security: Agricultural interventions are matched with field training for government sectors working with quilombolas communities on best agronomic practices to promote technical assistance for this communities. Stimulate the participation in the Program of Food Acquisition, supporting quilombolas agriculture.
  * For quilombolas participants: nutritional counseling based on traditional healthy cooking practices, using traditional recipes.
  * For health professionals: to strengthen food and nutrition actions at all levels of health care. Food and nutritional education training for primary care health professionals.
  * Helping families to have more knowledge about your citizen rights.
  Interventions: Other: Multi-sector interventions
- Control (Placebo Comparator): Conventional approach of current public food and nutrition policies.
  Interventions: Other: Control

INTERVENTIONS:
Other: Multi-sector interventions — * Multi-sector interventions to enhance food security: Agricultural interventions are matched with field training for government sectors working with quilombolas communities on best agronomic practices to promote technical assistance for this communities. Stimulate the participation in the Program of Food Acquisition, supporting quilombolas agriculture.
  * For quilombolas participants: nutritional counseling based on traditional healthy cooking practices, using traditional recipes.
  * For health professionals: to strengthen food and nutrition actions at all levels of health care. Food and nutritional education training for primary care health professionals.
  * Helping families to have more knowledge about your citizen rights.
  Arms: Multi-sector interventions
Other: Control — Placebo Comparator: Conventional approach of current public food and nutrition policies.
  Other Names: Placebo
  Arms: Control

SUMMARY:
To optimize the food security in quilombolas communities with high prevalence of food insecurity and obesity, the present study proposes to test a multi-sector intervention including agriculture sectors, health professionals and family members of communities, based on promotion of traditional food practices, health eating and enforceability of human right to adequate food.

DETAILED DESCRIPTION:
The present study proposes to develop nutrition education strategies through multi-sector intervention in order to promote the consumption of healthy foods and improvements in the health status of the quilombola population.This is a non-randomized cluster trial in four quilombolas communities in Southern Brazil (Passo do Lorenço, Algodão, Serrinha do Cristal and Nova Palma), combining qualitative and quantitative methodologies.

ELIGIBILITY:
Inclusion Criteria:

Quilombolas certified communities in Rio Grande do Sul, Brazil, with higher prevalence of food insecurity and obesity.

Exclusion Criteria:

Community leaders with no interest in study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Reduction in Brazilian Food Insecurity Scale score | 16 weeks after multisector intervention

SECONDARY OUTCOMES:
Improve consumption of healthy foods | 16 weeks after multisector intervention
  Healthy Eating Index (HEI) score. HEI is an indicator of dietary quality developed according to current Brazilian nutritional recommendations.
Number of participants who access food programs | 16 weeks after multisector intervention
Number of participants that improve knowledge about citizen rights. | 16 weeks after multisector intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marilda Neutzling, PhD, Principal Investigator — Post Graduate Studies Program in Epidemiology. Federal University of Rio Grande do Sul; Michele Drehmer, PhD, Study Chair — Post Graduate Studies Program in Epidemiology. Federal University of Rio Grande do Sul; Daniela Knauth, PhD, Study Chair — Post Graduate Studies Program in Epidemiology. Federal University of Rio Grande do Sul; Fernanda Bairros, PhD, Study Chair — Post Graduate Studies Program in Epidemiology. Federal University of Rio Grande do Sul
Locations (1):
- Pos-graduated Program in Epidemiology. Federal University of Rio Grande do Sul., Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Pacheco PM, Bairros FS, Neutzling MB, Nunes LN, Knauth DR, Dos Santos FS, Drehmer M. Effectiveness of a Nutrition Counseling Intervention on Food Consumption, According to the Degree of Processing: A Community-Based Non-Randomized Trial of Quilombola Communities in South Brazil. Int J Public Health. 2024 Nov 27;69:1607549. doi: 10.3389/ijph.2024.1607549. eCollection 2024. PMID 39664767